CLINICAL TRIAL: NCT04199364
Title: Comparison of Two Fraction Oxygen Inspired (FiO2) Thresholds for the Surfactant Administration in Preterm Infants With Respiratory Disease Syndrome: a Single-center Randomized Phase IV Clinical Trial
Brief Title: Medium vs Low Oxygen Threshold for the Surfactant Administration
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Virgilio Paolo Carnielli (Other)
Responsible Party: Sponsor-Investigator, Virgilio Paolo Carnielli, Director of Neonatology, Ospedali Riuniti Ancona
Organization: Ospedali Riuniti Ancona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2535; 2019-002923-13 (EudraCT Number)
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Distress Syndrome
Keywords: RDS; Surfactant; Threshold; Oxygen; Preterm; Infant
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth | interventions — poractant alfa

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low FiO2 threshold (Experimental): A fraction of inspired oxygen (FiO2) of 25% to have an oxygen saturation (SpO2) of 90-92%.
  Interventions: Drug: Poractant Alfa 80 mg/mL Intratracheal Suspension
- Medium FiO2 threshold (Experimental): A fraction of inspired oxygen (FiO2) of 35% to have an oxygen saturation (SpO2) of 90-92%.
  Interventions: Drug: Poractant Alfa 80 mg/mL Intratracheal Suspension

INTERVENTIONS:
Drug: Poractant Alfa 80 mg/mL Intratracheal Suspension — Exogenous surfactant (Poractant Alfa) administration at a dose of 200 mg/kg.

SUMMARY:
The aim of this study will be to assess the better fraction inspired oxygen (FiO2) threshold for the surfactant treatment in preterm infants with respiratory distress syndrome (RDS) randomized to receive exogenous surfactant at 25% or 35% of FiO2 threshold. The pulmonary gas-exchanges will be evaluated by oxygen saturation (SpO2) to FiO2 ratio (SFR) and will be used to define the better FiO2 threshold for the surfactant treatment.

DETAILED DESCRIPTION:
Exogenous surfactant therapy is an effective treatment of neonatal respiratory distress syndrome (RDS) and has been associated with reduced severity of respiratory distress and mortality. The 2019 European guidelines for neonatal RDS treatment suggest as the threshold of inspired oxygen (FiO2) for the surfactant treatment at 30% for all gestational age, but there are no randomized studies that confirm this indication. Some observational studies reported that a relevant number of patients who are not routinely treated with surfactant had respiratory complications, thus they received exogenous surfactant. To date, the optimal FiO2 threshold for surfactant administration remains unclear.

In this single-center, randomized, phase 4 trial, preterm infants (gestational age<32 weeks) with RDS will be randomized to receive exogenous surfactant at 25% or 35% of FiO2 threshold. According to the unit policy, the exogenous surfactant will be administered by an endotracheal tube in intubated infants, or by Intubation-Surfactant-Extubation (InSurE) / Less Invasive Surfactant Administration (LISA) methods in infants who will not remain intubated. The method used for the surfactant administration will be at the discretion of the caring physician.

ELIGIBILITY:
Inclusion Criteria:

* gestational age less than 32 weeks;
* diagnosis of respiratory distress (RDS);
* need for ventilatory support;
* written informed consent.

Exclusion Criteria:

* congenital malformations;
* genetic disorders;
* perinatal asphyxia.
* neonatal pneumonia or wet lung or meconium aspiration syndrome at birth.

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory pulmonary function | At day 3 of life
  The oxygen saturation (SpO2) to fraction of inspired oxygen (FiO2) ratio (SFR)

SECONDARY OUTCOMES:
Endotracheal intubation | At day 3, 7 and 28 of life, and at 36 weeks of postmenstrual age or at the discharge if it occurs first
  The need of endotracheal intubation after surfactant administration
Oxygen therapy | At day 3, 7 and 28 of life, and at 36 weeks of postmenstrual age or at the discharge if it occurs first
  The need of oxygen therapy
Respiratory Support-1 | At day 3, 7 and 28 of life, and at 36 weeks of postmenstrual age or at the discharge if it occurs first
  The need of respiratory support
Respiratory Support-1 | At day 3, 7 and 28 of life, and at 36 weeks of postmenstrual age or at the discharge if it occurs first
  Oxygenation index as indicator of the intensity of ventilatory
Respiratory severity-1 | At day 3, 7 and 28 of life, and at 36 weeks of postmenstrual age or at the discharge if it occurs first
  Silvermann score as secondary respiratory severity index
Respiratory severity-2 | At day 3, 7 and 28 of life, and at 36 weeks of postmenstrual age or at the discharge if it occurs first
  Lung ultrasound score (LUS) score as secondary respiratory severity index
Long-term respiratory pulmonary function | At day 7 and 28 of life, and at 36 weeks of postmenstrual age or at the discharge if it occurs first, and 1 year of corrected age
  The oxygen saturation (SpO2) to fraction of inspired oxygen (FiO2) ratio (SFR)
Complications of prematurity | From birth to 36 weeks of postmenstrual age or discharge if it occurred first
  The incidence of intraventricular hemorrhage of grade 3-4, periventricular leukomalacia, bronchopulmonary dysplasia, sepsis and retinopathy of prematurity
In-hospital death | From birth to 36 week of gestation or discharge if it occurred first
  death before 36 weeks of gestation

REFERENCES:
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2019 Update. Neonatology. 2019;115(4):432-450. doi: 10.1159/000499361. Epub 2019 Apr 11. PMID 30974433
- [Background] Engle WA; American Academy of Pediatrics Committee on Fetus and Newborn. Surfactant-replacement therapy for respiratory distress in the preterm and term neonate. Pediatrics. 2008 Feb;121(2):419-32. doi: 10.1542/peds.2007-3283. PMID 18245434
- [Background] Jobe AH. Pulmonary surfactant therapy. N Engl J Med. 1993 Mar 25;328(12):861-8. doi: 10.1056/NEJM199303253281208. No abstract available. PMID 8441430
- [Background] Ammari A, Suri M, Milisavljevic V, Sahni R, Bateman D, Sanocka U, Ruzal-Shapiro C, Wung JT, Polin RA. Variables associated with the early failure of nasal CPAP in very low birth weight infants. J Pediatr. 2005 Sep;147(3):341-7. doi: 10.1016/j.jpeds.2005.04.062. PMID 16182673
- [Background] Fuchs H, Lindner W, Leiprecht A, Mendler MR, Hummler HD. Predictors of early nasal CPAP failure and effects of various intubation criteria on the rate of mechanical ventilation in preterm infants of <29 weeks gestational age. Arch Dis Child Fetal Neonatal Ed. 2011 Sep;96(5):F343-7. doi: 10.1136/adc.2010.205898. Epub 2011 Jan 30. PMID 21278432
- [Background] Dargaville PA, Gerber A, Johansson S, De Paoli AG, Kamlin CO, Orsini F, Davis PG; Australian and New Zealand Neonatal Network. Incidence and Outcome of CPAP Failure in Preterm Infants. Pediatrics. 2016 Jul;138(1):e20153985. doi: 10.1542/peds.2015-3985. PMID 27365307
- [Background] Pillai MS, Sankar MJ, Mani K, Agarwal R, Paul VK, Deorari AK. Clinical prediction score for nasal CPAP failure in pre-term VLBW neonates with early onset respiratory distress. J Trop Pediatr. 2011 Aug;57(4):274-9. doi: 10.1093/tropej/fmq047. Epub 2010 Jun 16. PMID 20558382
- [Background] Dargaville PA, Aiyappan A, De Paoli AG, Dalton RG, Kuschel CA, Kamlin CO, Orsini F, Carlin JB, Davis PG. Continuous positive airway pressure failure in preterm infants: incidence, predictors and consequences. Neonatology. 2013;104(1):8-14. doi: 10.1159/000346460. Epub 2013 Apr 4. PMID 23595061
- [Background] De Jaegere AP, van der Lee JH, Cante C, van Kaam AH. Early prediction of nasal continuous positive airway pressure failure in preterm infants less than 30 weeks gestation. Acta Paediatr. 2012 Apr;101(4):374-9. doi: 10.1111/j.1651-2227.2011.02558.x. Epub 2012 Jan 9. PMID 22150698
- [Background] Rocha G, Flor-de-Lima F, Proenca E, Carvalho C, Quintas C, Martins T, Freitas A, Paz-Dias C, Silva A, Guimaraes H. Failure of early nasal continuous positive airway pressure in preterm infants of 26 to 30 weeks gestation. J Perinatol. 2013 Apr;33(4):297-301. doi: 10.1038/jp.2012.110. Epub 2012 Aug 30. PMID 22935774
- [Background] Gulczynska E, Szczapa T, Hozejowski R, Borszewska-Kornacka MK, Rutkowska M. Fraction of Inspired Oxygen as a Predictor of CPAP Failure in Preterm Infants with Respiratory Distress Syndrome: A Prospective Multicenter Study. Neonatology. 2019;116(2):171-178. doi: 10.1159/000499674. Epub 2019 May 21. PMID 31112987
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GH, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2016 Update. Neonatology. 2017;111(2):107-125. doi: 10.1159/000448985. Epub 2016 Sep 21. PMID 27649091
- [Background] Walsh BK, Daigle B, DiBlasi RM, Restrepo RD; American Association for Respiratory Care. AARC Clinical Practice Guideline. Surfactant replacement therapy: 2013. Respir Care. 2013 Feb;58(2):367-75. doi: 10.4187/respcare.02189. PMID 23359726
- [Background] McCord FB, Curstedt T, Halliday HL, McClure G, Reid MM, Robertson B. Surfactant treatment and incidence of intraventricular haemorrhage in severe respiratory distress syndrome. Arch Dis Child. 1988 Jan;63(1):10-6. doi: 10.1136/adc.63.1.10. PMID 3279916
- [Background] Narendran V, Donovan EF, Hoath SB, Akinbi HT, Steichen JJ, Jobe AH. Early bubble CPAP and outcomes in ELBW preterm infants. J Perinatol. 2003 Apr-May;23(3):195-9. doi: 10.1038/sj.jp.7210904. PMID 12732855
- [Background] Hedstrom AB, Gove NE, Mayock DE, Batra M. Performance of the Silverman Andersen Respiratory Severity Score in predicting PCO2 and respiratory support in newborns: a prospective cohort study. J Perinatol. 2018 May;38(5):505-511. doi: 10.1038/s41372-018-0049-3. Epub 2018 Feb 9. PMID 29426853
- [Background] Pang H, Zhang B, Shi J, Zang J, Qiu L. Diagnostic value of lung ultrasound in evaluating the severity of neonatal respiratory distress syndrome. Eur J Radiol. 2019 Jul;116:186-191. doi: 10.1016/j.ejrad.2019.05.004. Epub 2019 May 7. PMID 31153563
- [Background] Li L, Yang Q, Li L, Guan J, Liu Z, Han J, Chao Y, Wang Z, Yu X. [The value of lung ultrasound score on evaluating clinical severity and prognosis in patients with acute respiratory distress syndrome]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2015 Jul;27(7):579-84. doi: 10.3760/cma.j.issn.2095-4352.2015.07.008. Chinese. PMID 26138420
- [Background] Trachsel D, McCrindle BW, Nakagawa S, Bohn D. Oxygenation index predicts outcome in children with acute hypoxemic respiratory failure. Am J Respir Crit Care Med. 2005 Jul 15;172(2):206-11. doi: 10.1164/rccm.200405-625OC. Epub 2005 Apr 7. PMID 15817802